CLINICAL TRIAL: NCT03751839
Title: Microarchitecture, Bone Strength and Fracture Risk in Long-term Type 1 Diabetes
Acronym: BOLD-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Christian Meier (Other)
Collaborators: Insel Gruppe AG, University Hospital Bern (Other); University Hospital Schleswig-Holstein (Other); University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor-Investigator, Christian Meier, Prof. Dr. med. Christian Meier, University Hospital, Basel, Switzerland
Organization: University Hospital, Basel, Switzerland (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EKNZ 2018-01517
Record Dates: First submitted 2018-10-31; First posted 2018-11-23 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Absorptiometry, Photon

STUDY DESIGN:
Intervention Model Description: Identical diagnostic procedures will be performed in participants with type 1 diabetes and age- and sex-matched controls.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diagnostic (Experimental): The investigators will examine all participants in the same way by performing biochemical tests, clinical tests, osteodensitometry, HRQCT and HRpQCT measurements.
  Interventions: Diagnostic Test: Biochemical Tests; Diagnostic Test: Osteodensitometry; Diagnostic Test: Clinical Tests; Diagnostic Test: HR-QCT; Diagnostic Test: HR-pQCT

INTERVENTIONS:
Diagnostic Test: Biochemical Tests — The investigators will perform blood tests in every participant.
Diagnostic Test: Osteodensitometry — The investigators will perform an osteodensitometry in every participant.
  Other Names: dual energy x-ray absorptiometry (DXA scan)
Diagnostic Test: Clinical Tests — The investigators perform the following clinical tests: vibration threshold test, monofilament test, chair rise test and timed up and go test in every participant.
Diagnostic Test: HR-QCT — The investigators will perform HR-QCT measurements of the proximal femur and tibia in every participant.
Diagnostic Test: HR-pQCT — The investigators will perform HR-pQCT measurements of the distal radius and distal tibia in every participant.

SUMMARY:
This single center case control study will assess differences in bone structure between women and men with longstanding type 1 diabetes (diabetes duration>/= 25 years) and healthy controls.

DETAILED DESCRIPTION:
Based on a cross-sectional approach the investigators aim to assess microstructural, biomechanical and densitometric bone characteristics in patients with longstanding type 1 diabetes and age- and sex-matches controls. The investigators examine whether the presence of microvascular disease and/or poor diabetic control is associated with an altered bone microarchitecture and whether any such effect is independent of bone mineral density. Furthermore, the investigators aim to look into the relationship between an altered bone microarchitecture and advanced glycation end product (AGE) formation as well as biochemical markers of bone formation and bone turnover. The study aims to identify type 1 diabetic patients with high fracture risk by assessing the discriminatory power of parameters of cortical and trabecular microstructure measured via high resolution peripheral quantitative computed tomography (HR-pQCT) of the distal radius and tibia and high resolution quantitative computed tomography (HR-QCT) of the proximal femur and tibia with and without adjustment for bone density.

ELIGIBILITY:
Inclusion Criteria:

* women and men with longstanding type 1 diabetes (age 40-80 years, BMI 18-37 kg/m2 and age- and sex matched non-diabetic controls
* presence of type 1 diabetes for at least 25 years (defined by history of Insulin treatment)

Exclusion Criteria:

* Patients unable to give written informed consent, e.g. with severe dementia or patients not understanding German (or other local language)
* Any medical or psychiatric condition which would preclude the participant from adhering to the protocol
* Idiopathic or premenopausal osteoporosis or coexisting metabolic bone disease (e.g. Paget´s disease, primary hyperparathyroidism)
* Previous treatment with osteoporosis medication (bisphosphonates, denosumab) or intake of medications that are known to affect bone metabolism (e.g. steroids, anticonvulsants) within 6 months prior to enrollment
* Patients with medical conditions known to affect bone health ( e.g. metastatic bone disease, celiac disease, inflammatory bone disease, hypogonadism, thyrotoxicosis, hypercortisolism, chronic kidney disease stage IV and V (KDIGO), liver dysfunction (serum aspartate amino transferase (ASAT) >3 times the upper limit of normal)
* Inability to keep the extremities still for a few minutes of an HR-pQCT examination (e.g. Parkinson disease, spastic syndrome)
* Pregnant or breastfeeding women

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
volumetric bone mineral density in mg hydroxyapatite (HA)/ccm | through study completion, an average of 6 months
  measured by HR-pQCT at the distal radius and tibia
cortical porosity in % | through study completion, an average of 6 months
  measured by HR-pQCT at the distal radius and tibia
bone stiffness in kilonewton (kN)/mm | through study completion, an average of 6 months
  a measure of bone strength, measured by HR-pQCT at the distal radius and tibia
failure load in kN | through study completion, an average of 6 months
  a measure of bone strength, measured by HR-pQCT at the distal radius and tibia

SECONDARY OUTCOMES:
areal bone mineral density of the spine in g/cm2 | through study completion, an average of 6 months
  measured by osteodensitometry (DXA)
areal bone mineral density of the proximal femur in g/cm2 | through study completion, an average of 6 months
  measured by osteodensitometry
areal bone mineral density of the distal radius in g/cm2 | through study completion, an average of 6 months
  measured by osteodensitometry
trabecular bone score of the spine | through study completion, an average of 6 months
  a measure of bone texture, measured by osteodensitometry
cortical thickness at the mid tibia in cm | through study completion, an average of 6 months
  the cortical thickness will be measured by pulse-echo ultrasound and high resolution quantitative computed tomography (HR-QCT)
density weighed cortical thickness at the mid tibia in cm | through study completion, an average of 6 months
  the density weighed cortical thickness will be measured by pulse-echo ultrasound and HR- QCT
bone marrow adiposity in mg/cm3 | through study completion, an average of 6 months
  measured by HR-pQCT
measurement of serum carboxy-terminal collagen crosslinks (CTX) in pg/ml | through study completion, an average of 6 months
  biochemical marker of bone resorption
measurement of serum n-terminal procollagen type 1 (P1NP) in mcg/l | through study completion, an average of 6 months
  biochemical marker of bone formation
measurement of serum pentosidine in pmol/m | through study completion, an average of 6 months
  biochemical marker associated with bone fragility
measurement of serum carboxymethyl-lysine (CML) in pmol/ml | through study completion, an average of 6 months
  biochemical marker associated with bone fragility
measurement of serum insulin in mU/ml | through study completion, an average of 6 months
  biochemical marker associated with bone fragility
measurement of serum sclerostin in pg/ml | through study completion, an average of 6 months
  biochemical marker associated with bone fragility
measurement of serum adiponectin in ng/ml | through study completion, an average of 6 months
  biochemical marker associated with bone fragility
measurement of serum insulin like growth factor -1 (IGF1) in nM | through study completion, an average of 6 months
  biochemical marker associated with bone fragility
measurement of serum ultrasensitive c-reactive protein (usCRP) in mg/l | through study completion, an average of 6 months
  biochemical marker associated with bone fragility
measurement of serum interleukin 6 (IL6) in pg/ml | through study completion, an average of 6 months
  biochemical marker associated with bone fragility
measurement of serum periostin in ng/ml | through study completion, an average of 6 months
  biochemical marker associated with bone fragility

CONTACTS AND LOCATIONS:
Overall Officials: Christian Meier, Prof., Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- Department of Endocrinology, Diabetology and Metabolism, University Hospital Basel, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: No
In the informed consent document participants can choose whether they agree to the further use of their coded data and biochemical material for future research purposes.